CLINICAL TRIAL: NCT02862964
Title: Accuro Versus Traditional Landmark Palpation Technique to Determine Accurate Spinal Level for Procedures
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Mohamed Tiouririne, MD, Associate Professor, University of Virginia
Other Study IDs: 18684
Record Dates: First submitted 2016-05-03; First posted 2016-08-11 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Low Back Pain
Keywords: back pain
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- identify L4-5: Level marked as L4-5 using Accuro and palpation
  Interventions: Other: identify L4/L5

INTERVENTIONS:
Other: identify L4/L5 — * For each participant, a provider will first attempt to identify the L4/L5 space using the traditional technique of palpating the iliac crests to estimate spinal level. The provider will mark this space on the person's back with a single dot from a marking pen. The provider will then use the Accuro to again attempt to identify the L4/L5 interspace and mark this point with two dots.
  * The participant will then be taken into the fluoroscopy suite for their scheduled procedure a metal instrument will be laid on the skin at the interspace or interspaces that were marked using the palpation and Accuro techniques. Metal instruments show up on fluoroscopy, but the skin markers will not.
  * The anesthesiology attending in the fluoroscopy suite will then confirm the true interspace position of these marks under fluoroscopy performed for the standard of care procedure

SUMMARY:
Currently, at UVA, handheld ultrasound devices (like those used to view an unborn baby) are only two dimensional. The Accuro is a three dimensional handheld ultrasound device. This device uses sound waves to create pictures of the spine in three dimensions. This may allow the physician to view the spine in more detail for procedures such as spinal anesthesia and other diagnostic procedures.

The investigators aim to assess the benefit of using the Accuro versus traditional landmark palpation technique to determine accurate spinal level for procedures. Patients who undergo interventional pain procedure per standard care under fluoroscopy and require the presence of an anesthesia provider at the UVA Pain Management Clinic will be approached for enrollment.

Anesthesia Providers will first identify the L4/L5 space using the traditional technique of palpating the iliac crests to estimate spinal level, which will be marked with a single dot from a marking pen. The provider will then use the Accuro 3000 to identify the L4/L5 interspace and mark this point with two dots. Participants will then be taken into the fluoroscopy suite for their scheduled procedure. Since the skin marks will not show up on fluoroscopy, and metal instrument will be laid on the skin at the interspace or interspaces that were marked using the palpation and Accuro techniques. The anesthesiology attending provider in the fluoroscopy suite will then confirm the true interspace position of these marks under fluoroscopy. It will then be recorded how many spaces off the palpation and Accuro techniques are from the intended L4/L5 level.

DETAILED DESCRIPTION:
Patients who are undergoing any interventional pain procedure under fluoroscopy at the UVA Pain Management Clinic will be approached for consent.

* Each participant will sit up on the edge of the bed in the pre-procedural area of fluoroscopy.
* For each participant, a provider will first attempt to identify the L4/L5 space using the traditional technique of palpating the iliac crests to estimate spinal level. The provider will mark this space on the person's back with a single dot from a marking pen. The provider will then use the Accuro to again attempt to identify the L4/L5 interspace and mark this point with two dots.
* The participant will then be taken into the fluoroscopy suite for their scheduled procedure a metal instrument will be laid on the skin at the interspace or interspaces that were marked using the palpation and Accuro techniques. Metal instruments show up on fluoroscopy, but the skin markers will not.
* The anesthesiology attending in the fluoroscopy suite will then confirm the true interspace position of these marks under fluoroscopy performed for the standard of care procedure.
* The participant will not be exposed to any additional Fluro/ radiation time for this study
* It will then be recorded by the anesthesia provider, how many spaces off the palpation and Accuro techniques are from the intended L4/L5 level.

ELIGIBILITY:
Inclusion Criteria:

* An anesthesia provider under fluoroscopy at the UVA Pain Management Clinic

Exclusion Criteria:

* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing any interventional pain procedure requiring the presence of an anesthesia provider under fluoroscopy at the UVA Pain Management Clinic
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2016-02; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Accuracy in identifying the L4-L5 interspace using palpation versus ultrasound imaging (3D). | day one
  whether there is a correlation between the landmark traditional technique versus US imaging. Fluoroscopy will serve a s the control (gold standard)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Tiouririne, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin KJ, Perlas A, Chan V, Brown-Shreves D, Koshkin A, Vaishnav V. Ultrasound imaging facilitates spinal anesthesia in adults with difficult surface anatomic landmarks. Anesthesiology. 2011 Jul;115(1):94-101. doi: 10.1097/ALN.0b013e31821a8ad4. PMID 21572316
- [Background] Vallejo MC, Phelps AL, Singh S, Orebaugh SL, Sah N. Ultrasound decreases the failed labor epidural rate in resident trainees. Int J Obstet Anesth. 2010 Oct;19(4):373-8. doi: 10.1016/j.ijoa.2010.04.002. Epub 2010 Aug 8. PMID 20696564
- [Background] Grau T, Leipold RW, Conradi R, Martin E. Ultrasound control for presumed difficult epidural puncture. Acta Anaesthesiol Scand. 2001 Jul;45(6):766-71. doi: 10.1034/j.1399-6576.2001.045006766.x. PMID 11421838
- [Background] Grau T, Bartusseck E, Conradi R, Martin E, Motsch J. Ultrasound imaging improves learning curves in obstetric epidural anesthesia: a preliminary study. Can J Anaesth. 2003 Dec;50(10):1047-50. doi: 10.1007/BF03018371. PMID 14656785
- [Background] Chin KJ, Karmakar MK, Peng P. Ultrasonography of the adult thoracic and lumbar spine for central neuraxial blockade. Anesthesiology. 2011 Jun;114(6):1459-85. doi: 10.1097/ALN.0b013e318210f9f8. PMID 21422997